CLINICAL TRIAL: NCT00462969
Title: Cytologic Analysis of Distention Media as a Screening Test for Endometrial Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: American College of Obstetricians and Gynecologists (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CC06701; H-2006-0333 (Other: Health Sciences Institutional Review Board); NCI-2014-01355 (Registry Identifier: NCI Trial ID); A532820 (Other: UW Madison); SMPH\OBSTET & GYNECOL\ONC (Other: UW Madison); P30CA014520 (NIH)
Record Dates: First submitted 2007-04-17; First posted 2007-04-19 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2015-01

CONDITIONS: Endometrial Cancer
Keywords: Endometrial cancer; Sonohysterography
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): pre-surgical SHG
  Interventions: Procedure: Sonohysterography

INTERVENTIONS:
Procedure: Sonohysterography — Sonohysterography

SUMMARY:
The purpose of this study is to learn fluid from sonohysterography can be used to diagnose endometrial cancer.

DETAILED DESCRIPTION:
Participants will have a sonohysterography (SHG) performed. Fluid will be collected after instillation of 5mls of saline and again after an adequate SHG is performed. A pathologist will review this fluid to see is cancer cells are present.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed early-stage endometrial cancer

Exclusion Criteria:

* Recurrent or persistent endometrial cancer
* Evidence of distant metastases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Cytology results | At completion of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: David M Kushner, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- [Result] Guralp O, Sheridan SM, Harter J, Hinshaw JL, Seo S, Hartenbach EM, Lindheim S, Stewart S, Kushner DM. A new diagnostic test for endometrial cancer?: Cytology analysis of sonohysterography distention media. Int J Gynecol Cancer. 2013 Sep;23(7):1252-7. doi: 10.1097/IGC.0b013e31829fe8f6. PMID 23881100
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu